CLINICAL TRIAL: NCT04410614
Title: Dimensional Changes of Free Epithelial Graft at Teeth and Implant Sites: A Prospective Clinical Study
Brief Title: Dimensional Changes of Free Epithelial Graft at Teeth and Implant Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Principal Investigator, Alberto Monje, Head of Division of Periodontology, Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21052020
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Keratinized Mucosa
MeSH Terms: interventions — Chewing Gum; Transplantation

STUDY DESIGN:
Intervention Model Description: Teeth and implants receiving free epithelial grafts harvested from the palate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Free epithelial graft (Experimental): Free epithelial graft at implant and teeth sites to increase the band of keratinized mucosa
  Interventions: Procedure: Free epithelial (gingival) graft

INTERVENTIONS:
Procedure: Free epithelial (gingival) graft — 1mm thickness epithelial layer harvested from the palate (1st molar area) is grafted and stabilised at the dental or implant area deficient of keratinized mucosa

SUMMARY:
For the management of peridontal and peri-implant conditions, free epithelial grafts have been proposed to provide a sufficient band of keratinized mucosa with the goal of enhancing confort during brushing and reducing the level of inflammation. Nevertheless, these are subjected to dimensional changes that may jeopardise the final outcome of providing sufficient keratinized mucosa to teeth and implants. Hence, this prospective study will aim at shedding light on the dimensional changes and the variables affecting these changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of keratinized mucosa to improve the periodontal and peri-implant condition
* With no uncontrolled disease
* Non-smokers

Exclusion Criteria:

* Patients with uncontrolled diseases and conditions
* Smokers
* Patients with sufficient keratinized mucosa

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in keratinized mucosa | 3 weeks, 3 months, 6 months follow-up
  Area of keratinized mucosa gain

SECONDARY OUTCOMES:
Factor 1 affecting the dimensional changes | 3 weeks, 3 months, 6 months
  Avascular area exposed to the graft (implant/tooth surface)
Factor 2 affecting the dimensional changes | 3 weeks, 3 months, 6 months
  Thickness in mm of the graft
Factor 3 affecting the dimensional changes | 3 weeks, 3 months, 6 months
  Thickness in mm of the recipient connective tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Implantologia Cirugia Oral y Maxilofacial, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monje A, Blasi G. Significance of keratinized mucosa/gingiva on peri-implant and adjacent periodontal conditions in erratic maintenance compliers. J Periodontol. 2019 May;90(5):445-453. doi: 10.1002/JPER.18-0471. Epub 2018 Dec 7. PMID 30461016
- [Derived] Monje A, Blasi G, Amerio E, Sanz-Martin I, Nart J. Dimensional changes in free epithelialized gingival/mucosal grafts at tooth and implant sites: A prospective cohort study. J Periodontol. 2022 Jul;93(7):1014-1023. doi: 10.1002/JPER.21-0521. Epub 2022 Jan 25. PMID 34970744